CLINICAL TRIAL: NCT01054313
Title: A Phase I Trial of Docetaxel and Sirolimus in Patients With Advanced Malignancies
Brief Title: Docetaxel and Sirolimus in Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0558; NCI-2011-00545 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-01-20; First posted 2010-01-22 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Advanced Cancer
Keywords: Advanced Malignancies; Taxotere; Docetaxel; Rapamycin; Sirolimus; Rapamune; Prednisone; Resistant to standard therapy
MeSH Terms: interventions — Docetaxel; Sirolimus; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Docetaxel + Sirolimus (Experimental): Starting doses of Docetaxel 30 mg/m^2 IV every 3 weeks + Sirolimus 1 mg daily
  Interventions: Drug: Docetaxel (Taxotere); Drug: Sirolimus (Rapamycin); Drug: Prednisone

INTERVENTIONS:
Drug: Docetaxel (Taxotere) — Starting dose 30 mg/m^2 by vein (IV) over about 1 hour on Day 1 of every 21 day cycle.
Drug: Sirolimus (Rapamycin) — Starting dose 1 mg daily by mouth 1 time a day.
  Other Names: Rapamune
Drug: Prednisone — 5 mg by mouth twice a day with prostate cancer.

SUMMARY:
The goal of this clinical research study to find the highest tolerated dose of the combination of Taxotere (docetaxel) and Rapamycin (sirolimus) when given to patients with advanced cancer.

Researchers also want to find highest tolerated dose of the combination of docetaxel, sirolimus, and prednisone when given to patients with advanced prostate cancer. The safety of both drug combinations will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Docetaxel is designed to stop the growth of cancer cells, which may cause the cells to die. It is believed to be weakly effective at killing blood vessels in tumor tissue as well.

Sirolimus is designed to block a protein called mammalian target of rapamycin (mTOR) inside the cancer cell.

Prednisone is a corticosteroid that is similar to a natural hormone made by your body. Prednisone is often given in combination with chemotherapy to treat cancer.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of the combination of docetaxel and sirolimus based on when you joined this study. Up to 12 dose levels of docetaxel and sirolimus will be tested. Three (3) to 6 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of docetaxel and sirolimus is found. Once the highest tolerable dose of docetaxel and sirolimus is found, up to 12 more patients may be enrolled to further study the safety of the drug at each of that dose.

If you have prostate cancer, you will also receive prednisone. All participants who receive prednisone will receive the same dose level.

Study Drug Administration:

Each study cycle is 21 days.

Everyday, you will take sirolimus by mouth 1 time a day. Sirolimus can be taken with or without food, but should be taken at the same time everyday.

On Day 1 of every cycle, you will receive docetaxel by vein over about 1 hour.

If you are taking prednisone, you will take it 2 times every day by mouth with food and water.

Study Visits:

Every week for the first 3 weeks and then about every 3 weeks, blood (about 5 teaspoons) will be drawn for routine tests. You will also have a physical exam.

Every 6 weeks, women who are able to have children will have blood drawn for a pregnancy test.

About every three weeks, blood (about 5 teaspoons) will be drawn for routine tests, to check your kidney function, and for biomarker tests.

About every 6 weeks, you will have a CT scan and x-ray to check the status of the disease.

Length of Study:

You will be on study for as long as you are benefitting. You will be taken off the study if the disease gets worse or you experience intolerable side effects.

Follow-Up:

If you experience intolerable side effects, you will be followed until the side effect has resolved or the side effect does not continue to improve or get worse. The study doctor will tell you what tests will need to be performed.

This is an investigational study. Docetaxel is FDA approved and commercially available for the treatment of advanced cancers such as breast, lung, and prostate cancer. Sirolimus is FDA approved and commercially available for the prevention of transplant rejection in kidney transplant patients. Prednisone is FDA approved and commercially available for the treatment of prostate cancer when given with docetaxel.

The combination of docetaxel and sirolimus, with or without prednisone, to treat advanced cancer is investigational. Most patients in this study will receive docetaxel and sirolimus. However, if you have prostate cancer, you will receive docetaxel, prednisone, and sirolimus.

Up to 68 patients will be enrolled in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced or metastatic cancer that is refractory to standard therapy, relapsed after standard therapy, or who have no standard therapy available that improves survival by at least three months.
2. Patients must be at least 5 half-lives or three weeks, whichever is shorter, from their previous targeted or biologic therapy; patients must be at least three weeks beyond previous cytotoxic therapy. In addition, patients must be >/= 3 weeks beyond previous therapeutic radiation or major surgery. Patients may have received palliative localized radiation immediately before or during treatment providing radiation is not delivered only to the site of disease being treated under this protocol. Terminal phase half life of docetaxel is 11.1 hours; sirolimus, 14.5 hours.
3. cont'd from criterion #2 Previous mTOR inhibitor (everolimus, temsirolimus, and sirolimus) and taxane (including paclitaxel, abraxane/ABI-007, and docetaxel) therapy is permitted.
4. Eastern Cooperative Oncology Group (ECOG) performance status </= 3
5. Patients must have normal organ and marrow function defined as:absolute neutrophil count >/= 1,000/mL; platelets >/=50,000/mL; creatinine </= 2 x upper limit of normal (ULN); total bilirubin </= 3x ULN; ALT(SGPT) </= 3 x ULN; cholesterol </= 350 mg/dL; triglycerides </= 400 mg/dL.
6. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 30 days after the last dose.
7. Patients must be able to understand and be willing to sign a written informed consent document.
8. Patients already on gonadotropin-releasing hormone (GnRH) agonist therapy (eg goserelin acetate, leuprolide acetate) for metastatic, castrate-resistant prostate cancer for three months prior to entry into this study may be continued on this intervention while enrolled in this protocol. Patients on somatostatin analogues (eg octreotide) for symptom control for three months prior to entry into this study may be continued on this intervention while enrolled in this protocol.

Exclusion Criteria:

1. Uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, uncontrolled asthma, need for hemodialysis, and need for ventilatory support.
2. Pregnant or lactating women.
3. History of hypersensitivity to docetaxel or any component of the formulation.
4. History of hypersensitivity to sirolimus or any component of the formulation
5. Patients maintained on medications that are strong inducers or inhibitors of CYP3A4 should have these medications discontinued prior to entry on study unless cessation of such medications would be detrimental to patient's health.
6. Patients unwilling or unable to sign informed consent document.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2010-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose(MTDs) for Docetaxel - Sirolimus | Every week for first 3 weeks then every 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Filip Janku, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org